CLINICAL TRIAL: NCT04312789
Title: A Phase II Trial of Avatrombopag for the Treatment of Thrombocytopenia After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Avatrombopag for the Treatment of Thrombocytopenia After Donor Hematopoietic Stem Cell Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug availability
Sponsor: Ayman Saad (Other)
Collaborators: Sobi, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ayman Saad, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19328; NCI-2020-01035 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Platelet Disorder
MeSH Terms: conditions — Blood Platelet Disorders | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (avatrombopag) (Experimental): Patients receive avatrombopag PO QD for up to 1 year in the absence of disease progression or unacceptable toxicity. Avatrombopag will be titrated weekly until platelet count of greater than or equal to 60,000/uL is achieved and persists for 7 consecutive days, and the patient remains free from platelet transfusion.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — Given PO
  Other Names: AKR-501; AS 1670542; Doptelet; E5501; YM 477

SUMMARY:
This phase II trial studies the side effects and how well avatrombopag works for the treatment of thrombocytopenia after donor hematopoietic stem cell transplant. Thrombocytopenia is defined as abnormally low level of platelets in the blood. Avatrombopag is a small molecule thrombopoietin receptor agonist which stimulates thrombopoietin receptor leading to increase production of platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and efficacy of avatrombopag for the treatment of thrombocytopenia after allogenic hematopoietic stem cell transplantation.

SECONDARY OBJECTIVE:

I. To identify predictors of response to avatrombopag.

OUTLINE:

Patients receive avatrombopag orally (PO) once daily (QD) for up to 1 year in the absence of disease progression or unacceptable toxicity. Avatrombopag will be titrated weekly until platelet count of greater than or equal to 60,000/uL is achieved and persists for 7 consecutive days, and the patient remains free from platelet transfusion.

After completion of study treatment, patients are followed up weekly for 4 weeks and then monthly up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Failure to engraft platelets by day 30 (D30) after hematopoietic cell transplantation (HCT) defined as: Platelet count less than 20,000/uL and patient is still dependent on platelet transfusion support
* Patient must be able to start treatment with avatrombopag within 30-60 days following transplant
* Able to provide written informed consent from patient or legal representative

Exclusion Criteria:

* Serious uncontrolled infections
* Steroid refractory graft versus host disease (GVHD)
* Patients with thrombotic microangiopathy
* Pregnant or lactating women
* Creatinine clearance < 30 ml/min
* Active thromboembolism requiring anticoagulation
* Unable to understand the investigational nature of the study or provide informed consent
* Evidence of disease relapse by flow cytometry of chimerisms
* Concomitant use of other thrombopoietin receptor agonists (TPO-RA) medication during the treatment phase of the study or two weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events of avatrombopag treatment | Up to 30 days after the last dose
  Toxicities will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version (v).5 standard toxicity grading. Frequency and other descriptive statistics will be used to present the toxicity pattern.
Failure rate of platelet recovery | At day 90
  The proportion will be provided with 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Independence from platelet transfusion | Up to 1 year
Duration of platelet response | Up to 1 year
  Will be presented in a descriptive manner.
Platelet count >= 50,000/uL for 7 consecutive days without transfusion support | Up to 1 year
Duration of exposure to avatrombopag | Up to 1 year
  Will be presented in a descriptive manner.
Incidence of adverse events associated with avatrombopag treatment | Up to 30 days after last dose
Transplant-related mortality | At day 100 and 1 year post-hematopoietic stem cell transplant (HCT)
Progression-free survival (PFS) of underlying malignant hematologic disorder | From the time of HCT to progression and death, assessed up to 1 year
  The method of Kaplan-Meier will be used to estimate PFS.
Overall survival (OS) | From the time of HCT to death from any cause, assessed up to 1 year
  The method of Kaplan-Meier will be used to estimate OS.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Saad, MB/BCH, Principal Investigator — Ohio State University Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu